CLINICAL TRIAL: NCT04328961
Title: Efficacy of Hydroxychloroquine for Post-exposure Prophylaxis (PEP) to Prevent Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection Among Adults Exposed to Coronavirus Disease (COVID-19): a Blinded, Randomized Study
Brief Title: Hydroxychloroquine for COVID-19 Post-exposure Prophylaxis (PEP)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Ruanne Barnabas, Associate Professor, School of Medicine: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00009750; INV-016204 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2020-03-23; First posted 2020-04-01 (Actual); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Corona Virus Infection; SARS (Severe Acute Respiratory Syndrome); SARS-CoV-2
Keywords: novel coronavirus; post-exposure prophylaxis
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — Hydroxychloroquine; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ascorbic Acid (Placebo Comparator): Ascorbic acid 500 mg orally daily for 3 days, then 250 mg orally daily for 11 days
  Interventions: Drug: Ascorbic Acid
- Hydroxychloroquine (Experimental): Hydrochloroquine 400 mg orally daily for 3 days, then 200 mg orally daily for an additional 11 days
  Interventions: Drug: Hydroxychloroquine Sulfate

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — Eligible participants in a household randomized to this study arm will receive hydrochloroquine therapy
  Other Names: HCQ arm
  Arms: Hydroxychloroquine
Drug: Ascorbic Acid — Eligible participants in a household randomized to this study arm will receive ascorbic acid therapy.
  Other Names: Placebo arm
  Arms: Ascorbic Acid

SUMMARY:
This is a clinical study for the prevention of SARS-CoV-2 infection in adults exposed to the virus. This study will enroll up to 2000 asymptomatic men and women 18 to 80 years of age (inclusive) who are close contacts of persons with laboratory confirmed SARS-CoV-2 or clinically suspected COVID-19. Eligible participants will be enrolled and randomized to receive the intervention or placebo at the level of the household (all eligible participants in one household will receive the same intervention).

DETAILED DESCRIPTION:
This is a randomized, multi-center, placebo-equivalent (ascorbic acid) controlled, blinded study of Hydroxychloroquine (HCQ) post-exposure prophylaxis (PEP) for the prevention of SARS-CoV-2 infection in adults exposed to the virus.The overarching goal of this study is to assess the effectiveness of HCQ PEP on the incidence of SARS-CoV-2 detection by polymerase chain reaction (PCR) to inform public health control strategies.This study will enroll up to 2000 asymptomatic men and women 18 to 80 years of age (inclusive) at baseline who are close contacts of persons with PCR-confirmed SARS-CoV-2 or clinically suspected COVID-19 and a pending SARS-CoV-2 PCR test. Eligible participants will be enrolled and randomized 1:1 to HCQ or ascorbic acid at the level of the household (all eligible participants in one household will receive the same intervention). Participants will be counseled about the preliminary in vitro data on HCQ activity against SARS CoV-2 and equipoise regarding efficacy in humans.The duration of study participation will be approximately 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 80 years of age inclusive, at the time of signing the informed consent
* Willing and able to provide informed consent
* Had a close contact of a person (index) with known PCR-confirmed SARS-CoV-2 infection or who is currently being assessed for COVID-19. Close contact defined as:

  1. Household contact (i.e., residing with the index case in the 14 days prior to index diagnosis)
  2. Medical staff, first responders, or other care persons who cared for the index case without personal protection (mask and gloves)
* Less than 4 days since last exposure (close contact with a person with SARS-CoV-2 infection) to the index case
* Body weight < 100 kg (self-reported)
* Access to device and internet for Telehealth visits

Exclusion Criteria:

* Known hypersensitivity to HCQ or other 4-aminoquinoline compounds
* Currently hospitalized
* Symptomatic with subjective fever, cough, or sore throat
* Current medications exclude concomitant use of HCQ
* Concomitant use of other anti-malarial treatment or chemoprophylaxis
* History of retinopathy of any etiology
* Psoriasis
* Porphyria
* Known bone marrow disorders with significant neutropenia (polymorphonuclear leukocytes < 1500) or thrombocytopenia (< 100 K)
* Concomitant use of digoxin, cyclosporin, cimetidine, or tamoxifen
* Known liver disease
* Known long QT syndrome
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of the study drugs, or planned use during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 943 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne V. Barnabas, MBChB, DPhil, Principal Investigator — University of Washington
Locations (8):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - Tulane, New Orleans, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Washington, Coordinating Center, Seattle, Washington
  - UW Virology Research Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the study will be made available in accordance with the funder's open access policy.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Within 3 months of publication of primary results.
Access Criteria: De-identified data from the study will be made available in accordance with the funder's open access policy.
URL: https://www.gatesfoundation.org/how-we-work/general-information/open-access-policy

REFERENCES:
- [Derived] Barnabas RV, Brown ER, Bershteyn A, Stankiewicz Karita HC, Johnston C, Thorpe LE, Kottkamp A, Neuzil KM, Laufer MK, Deming M, Paasche-Orlow MK, Kissinger PJ, Luk A, Paolino K, Landovitz RJ, Hoffman R, Schaafsma TT, Krows ML, Thomas KK, Morrison S, Haugen HS, Kidoguchi L, Wener M, Greninger AL, Huang ML, Jerome KR, Wald A, Celum C, Chu HY, Baeten JM; Hydroxychloroquine COVID-19 PEP Study Team. Hydroxychloroquine as Postexposure Prophylaxis to Prevent Severe Acute Respiratory Syndrome Coronavirus 2 Infection : A Randomized Trial. Ann Intern Med. 2021 Mar;174(3):344-352. doi: 10.7326/M20-6519. Epub 2020 Dec 8. PMID 33284679
- [Derived] Barnabas RV, Brown E, Bershteyn A, Miller RS, Wener M, Celum C, Wald A, Chu H, Wesche D, Baeten JM; Hydroxychloroquine COVID-19 PEP Study Team. Efficacy of hydroxychloroquine for post-exposure prophylaxis to prevent severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection among adults exposed to coronavirus disease (COVID-19): a structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 3;21(1):475. doi: 10.1186/s13063-020-04446-4. PMID 32493478

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 949 participants were assessed for eligibility, 114 were excluded and 829 were randomized.
Period: Overall Study
Arm/Group | Ascorbic Acid | Hydroxychloroquine
Started | 422 | 407
Completed | 336 | 353
Not Completed | 86 | 54

BASELINE CHARACTERISTICS:
Population: The above participants contributed to the Modified Intention-to-Treat Cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ascorbic Acid | Hydroxychloroquine | Total
Number analyzed (Participants) | 336 | 353 | 689
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 307 | 322 | 629
  >=65 years | 29 | 31 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 38 [26 to 50] | 40 [27 to 51] | 39 [27 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 215 | 412
  Male | 139 | 138 | 277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 86 | 69 | 155
  Not Hispanic or Latino | 250 | 284 | 534
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 7 | 12
  Asian | 43 | 30 | 73
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 34 | 20 | 54
  White | 160 | 209 | 369
  More than one race | 86 | 69 | 155
  Unknown or Not Reported | 7 | 17 | 24
Region of Enrollment [Number; unit: participants]
  United States | 336 | 353 | 689

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Polymerase Chain Reaction (PCR) Confirmed SARS-CoV-2 Infection
Description: Polymerase chain reaction (PCR) confirmed severe acute respiratory syndrome coronavirus 2 of the genus Betacoronavirus (SARS-CoV-2) infection from self-collected samples collected daily for 14 days
Time Frame: Day 1 through Day 14 after enrolment
Population: The above participants qualified for the Modified Intention-to-Treat Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Ascorbic Acid | Hydroxychloroquine
Number analyzed (Participants) | 336 | 353
Participants | 45 | 53

2. Primary Outcome: The Number of Participants Who Had Polymerase Chain Reaction (PCR) Confirmed SARS-CoV-2 Infection
Description: Polymerase chain reaction (PCR) confirmed SARS-CoV-2 infection from self-collected samples collected at study exit
Time Frame: Day 28 after enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Ascorbic Acid | Hydroxychloroquine
Number analyzed (Participants) | 336 | 353
Participants | 48 | 58

3. Secondary Outcome: Rate of Participant-reported Adverse Events
Description: Safety and tolerability of Hydroxychloroquine as SARS-CoV-2 PEP in adults
Time Frame: 28 days from start of Hydroxychloroquine therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Ascorbic Acid | Hydroxychloroquine
Number analyzed (Participants) | 336 | 353
Participants | 46 | 66

4. Secondary Outcome: Number of Participants Who Had COVID-19 Disease
Description: Participants who had a PCR-confirmed SARS-CoV-2 infection and met the Center for Disease Control (CDC) defined criteria for symptomatic COVID-19 disease.
Time Frame: 28 days from enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Ascorbic Acid | Hydroxychloroquine
Number analyzed (Participants) | 336 | 353
Participants | 26 | 37

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the period of follow up, which was 28 days.
Description: Adverse event collection was obtained through daily surveys completed by participants. If participants were experiencing symptoms they were contacted by study staff for more information.
Arm/Group | Ascorbic Acid | Hydroxychloroquine
All-Cause Mortality (participants affected / at risk) | 0/422 | 0/407
Serious Adverse Events (participants affected / at risk) | 2/422 | 2/407
Other Adverse Events (participants affected / at risk) | 46/422 | 66/407
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid (N=422) | Hydroxychloroquine (N=407)
Hospitalizations (Infections and infestations) | 1 (1) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid (N=422) | Hydroxychloroquine (N=407)
Diarrhea, abdominal discomfort, or vomiting (Gastrointestinal disorders) | 7 (7) | 25 (25)
Nausea or upset stomach (Gastrointestinal disorders) | 10 (10) | 14 (14)
Skin reaction/rash (Skin and subcutaneous tissue disorders) | 8 (8) | 11 (11)
Neurologic reaction: irritability, dizziness, or vertifgo (General disorders) | 11 (11) | 6 (6)
Headache (General disorders) | 7 (7) | 5 (5)
Hot flashes, night sweats, or palpitations (General disorders) | 6 (6) | 2 (2)
Taste change or dry mouth (General disorders) | 6 (6) | 1 (1)
Fatigue (General disorders) | 2 (2) | 4 (4)
Visual Changes (Eye disorders) | 0 (0) | 4 (4)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT04328961/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT04328961/SAP_001.pdf